CLINICAL TRIAL: NCT04880252
Title: In Individuals With Subjective Cognitive Decline, Age, Memory and Action Speed Scores at Baseline Predict Progression to Cognitive Impairment
Brief Title: Neuropsychological Indicators of SCD Progression
Acronym: SCD-CI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0039
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Biomarkers; Cognitive Assessment; Cognitive Decline; Neurocognitive Disorders; Neurodegenerative Diseases; Subjective Cognitive Decline
Keywords: Biomarkers; Cognitive assessment; Cognitive decline; Neurocognitive disorders; Neurodegenerative diseases; Neuropsychological assessment; Risk of progression; Subjective cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some patients with subjective cognitive decline (SCD) progress to neurocognitive disorders (NCD), whereas others remain stable; however, the neuropsychological determinants of this progression have not been identified. The investigators objective was to examine baseline neuropsychological indicators that could discriminate between people in whom the SCD progressed to a mild or major NCD and people in whom the SCD remained stable.

The investigators retrospectively included patients consulting for SCD at a university medical center's memory center (Amiens, France) and who had undergone three or more neuropsychological assessments at least 6 months apart. The relationship between domain-specific scores and the global cognitive score (GCS, as a function of final status (stable SCD vs. progression toward a mild or major NCD)) was examined using a generalized linear mixed model.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been referred to the memory center at Amiens University Medical Center (Amiens, France).
* patients who had undergone three neuropsychological assessments at least 6 months apart, from 2005
* patients who met the criteria for SCD.

Exclusion Criteria:

* patients who didn't meet the criteria for SCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for SCD at a university medical center's memory center (Amiens, France) and who had undergone three or more neuropsychological assessments at least 6 months apart.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Variation of neuropsychological indicators (global congnitive score) between NCD et SCD patients | one year
  subjective cognitive decline (SCD) neurocognitive disorders (NCD) neuropsychological indicators could discriminate between people in whom SCD progressed to a mild or major NCD and people in whom SCD remained stable.
  A global cognitive score was created using all 5 tests : Alice Heim 4-I tests inductive reasoning ; Short-term verbal memory was assessed with a 20-word free-recall test; Two measures of verbal fluency were used: phonemic and semantic; Vocabulary was assessed using the Mill Hill Vocabulary test.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perron A, Roussel M, Wannepain-Despretz S, Barbay M, Devendeville A, Godefroy O, Andriuta D. In Individuals With Subjective Cognitive Decline, Age, Memory and Speed Scores at Baseline Predict Progression to Cognitive Impairment. Alzheimer Dis Assoc Disord. 2022 Oct-Dec 01;36(4):359-361. doi: 10.1097/WAD.0000000000000520. Epub 2022 Jul 19. PMID 35867966